CLINICAL TRIAL: NCT06934057
Title: Cabozantinib and Nivolumab Among Older Patients With Renal-cell Carcinoma, a Prospective Cohort With Geriatric, Pharmacologic and Patient-reported-outcome Evaluation
Brief Title: Cabozantinib and Nivolumab Among Older Patients With Renal Cell Carcinoma
Acronym: CABOLD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516650-22-00; 2024/3873 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Kidney Cancer; Renal Cell Cancer
Keywords: renal cell carcinoma; kidney cancer; cabozantinib; nivolumab; elderly patients; geriatric population
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib-Nivolumab (Experimental): The patient will be treated according to standard of care Nivolumab Cabozantinib.
  Interventions: Drug: Nivolumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Nivolumab — Briefly, nivolumab is administered as an approximately 30-minute (240mg every 2 weeks) or 60-minute (480mg every 4 weeks) IV infusion.
  Other Names: OPDIVO
Drug: Cabozantinib — Cabozantinib is a medication that is taken orally every day, once a day away from meals at the initial dose of 40 mg/day.
  Other Names: CABOMETYX

SUMMARY:
The goal of the study is to describe real-life use and exposition to nivolumab-cabozantinib among older patients with metastatic clear-cell renal cell cancer

DETAILED DESCRIPTION:
This study will be a prospective, multicentric, single-arm cohort. Patients will receive Nivolumab-Cabozantinib association per standard. All patients will benefit of geriatric evaluation (G-CODE) at inclusion, and a multimodal and reinforced follow-up, including medical oncologist, geriatrician nurse of doctor, phone calls, and optional pharmacological follow-up for Cabozantinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 70 years-old
2. Confirmed advanced or metastatic renal-cell carcinoma
3. Patients not previously treated in metastatic setting
4. Performance Status 0 to 2
5. Sexually active male patients must agree to use condom during the study and for at least 5 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.
6. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
7. Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last four weeks and while on study treatment (Patients may be included in CABOLD if they are included in the arm B of CARE1 study EUCT N° 2023-503317-29-00)
2. Performance Status > 2
3. Any condition that represent a contraindication to Cabozantinib and/or Nivolumab, as described in summaries of products characteristics, including symptomatic untreated brain metastasis or active auto-immune disease requiring systemic immunosuppressant/modulator (thyroid or adrenal disorder are not an exclusion criteria)
4. Any severe cardiovascular or thrombo-embolic event in the last three months
5. Any situation for which exclusive palliative care intervention is recommended
6. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Starting dose of Cabozantinib | 24 weeks after treatment start
  Primary outcome measure is treatment patterns, which includes starting dose of cabozantinib.
Dose interruption of Cabozantinib | 24 weeks after treatment start
  Primary outcome measure is treatment patterns of Cabozantinib, which includes the proportion of patients who experience any temporary dose interruption within the first 24 weeks of treatment.
Dose modifications of Cabozantinib | 24 weeks after treatment start
  Primary outcome measure is treatment patterns, which includes the proportion of patients who experience any form of dose modification of Cabozantinib related to all grade toxicity within the first 24 weeks of treatment.

SECONDARY OUTCOMES:
Overall response rate based on radiological evaluation | 12 months after treatment start
  Overall response rate based on best radiological response rate with local RECIST 1.1 evaluation observed in the 12 months of the study
Overall-survival | 12 months after treatment start
  Defined as the time between the date of inclusion and the date of death whatever the cause. Patients alive at the date of last follow-up visit will be censored at that date.
Progression free survival | 12 months after treatment start
  Progression free survival, defined by the time between inclusion date and the date of observation of a progression of the disease according to RECIST 1.1 or death of the patient (all causes combined) or date of last follow-up if the patient is alive without progression or lost to follow up.
Duration of response | 12 months after treatment start
  It is defined as the time from first radiological evidence of response (partial or complete response) to disease progression or death among patients who achieve complete or partial response.
Frequency of adverse events according to CTCAE V5 | 12 months after treatment start
  Tolerance is evaluated based on physicians reports.
Frequency of adverse events according to PRO-CTCAE | 12 months after treatment start
  Tolerance is evaluated based on patients reports.
Quality of life - Patient-related outcomes - FACT-G | At baseline, and every 3 months after treatment start, up to 12 months after treatment start
  Patients reported quality of life is evaluated based on Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. It is an 27 item questionnaire, ranging from 0 to 108 score. Higher scores indicate better quality of life
Quality of life - Patient-related outcomes - FACIT TS-G | Every 3 months after treatment start, up to 12 months after treatment start
  Patients reported quality of life is evaluated based on Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT TS-G) questionnaire. The score range goes from 0 to 70 score. Higher scores indicate greater satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maxime FRELAUT, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (7):
- France (7):
  - Institut de Cancérologie de l'Ouest - Angers, Angers
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital Tenon, Paris
  - Institut Universitaire Du Cancer Toulouse- Oncopole Claudius Regaud, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No